CLINICAL TRIAL: NCT01106001
Title: A Double Blind Randomized Control Trial on the Efficacy of Periarticular Levo Bupivicaine Injection Following Primary Hip Arthroplasty
Brief Title: Study to Test the Efficacy of Periarticular Levo Bupivicaine Injection Following Primary Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orthopaedic Research and Innovation Foundation, Ireland (Other)
Responsible Party: Prof Kevin Mulhall, Orthopaedic Research and Innovation Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KM-042008-014
Record Dates: First submitted 2010-04-12; First posted 2010-04-19 (Estimated); Last update posted 2010-04-19 (Estimated); Status verified 2008-07

CONDITIONS: Osteoarthritis
Keywords: total hip arthroplasty; periarticular injection; pain
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Levobupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levobupivacaine (Active Comparator): Levobupivacaine is indicated for local anaesthesia including infiltration, nerve block, ophthalmic, epidural and intrathecal anaesthesia in adults; and infiltration analgesia in children
  Interventions: Drug: Levobupivacaine
- Saline (Placebo Comparator): Saline (also saline solution) is a general term referring to a sterile solution of sodium chloride (NaCl, more commonly known as salt) in water but is only sterile when it is placed intravenously, otherwise, a saline solution is a salt water solution.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Levobupivacaine — The treatment group received 150mg of levobupivicaine in 60mls of 0.9% saline. This was injected intra-operatively through the medial and anterior capsular spaces in the region of the obturator and femoral nerves and also around the short rotators and gluteus maximus in the region of the inferior and superior gluteal nerves. The timing of this was after insertion of the acetabular component. 10mls was then infiltrated around the tensor fascia lata and subcutaneously prior to closing the wound.
  Arms: Levobupivacaine
Drug: Saline — The placebo group received 60mls of 0.9% saline injected intra-operatively through the medial and anterior capsular spaces in the region of the obturator and femoral nerves and also around the short rotators and gluteus maximus in the region of the inferior and superior gluteal nerves. The timing of this was after insertion of the acetabular component. 10mls was then infiltrated around the tensor fascia lata and subcutaneously prior to closing the wound.
  Arms: Saline

SUMMARY:
The hypothesis of this study is that isolated use of local periarticular levobupivicaine injection during primary hip arthroplasty would improve post-operative pain control. Patients were randomised in the operating room to receive either a periarticular infiltration, or a placebo consisting of Saline. Morphine and analgesic consumption was recorded for each patient, while the modified McGill pain scale was used to determine the adequacy of analgesia and the benefit of the peri-articular infiltration. 91 patients were recruited, with 45 patients in the treatment group and 46 controls. The results were assessed after one year, once all the information from both treatment groups was collected.

DETAILED DESCRIPTION:
The efficacy of periarticular injections during total knee arthroplasty is well established but there is little published data on their effect in primary hip arthroplasty. We hypothesized that isolated use of local periarticular levobupivicaine injection during primary hip arthroplasty would improve post-operative pain control. A double blinded, randomised, placebo-controlled trial on patients undergoing primary hip arthroplasty was performed. Patients were randomised in theatre to receive either a periarticular infiltration of 150mg levobupivicaine in 60mls of 0.9% Saline, or a placebo consisting of 60mls 0.9% Saline. Morphine and analgesic consumption was recorded for each patient, while the modified McGill pain scale was used to determine the adequacy of analgesia and the benefit of the peri-articular infiltration. 91 patients were recruited, with 45 patients in the treatment group and 46 controls. The results were assessed after one year, once all the information from both treatment groups was collected.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing primary hip arthroplasty for osteoarthritis only were included in this study after giving informed consent.

Exclusion Criteria:

* Patients with cognitive impairment, neurological disorders, advanced liver or renal impairment, known ischemic heart disease, a previous diagnosis of a pain syndrome or any post-operative surgical or medical complications were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine a significant difference (p>0.05) in morphine consumption between the two treatment groups post-operatively. | 1 year
  The modified McGill pain scale was administered to determine the adequacy of analgesia and the benefit of the peri-articular infiltration. In addition, morphine and analgesic consumption was recorded for each patient. The results were assessed after one year, once all the information from both treatment groups was collected.

SECONDARY OUTCOMES:
To analyse the length of stay for between both treatment groups | Average 6 days (based on precise day of discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Mulhall, Principal Investigator — Orthopaedic Research and Innovation Foundation, Ireland
Locations (2):
- Ireland (2):
  - Cappagh National Orthopaedic Hospital, Dublin, Finglas
  - Orthopaedic Research and Innovation Foundation, Dublin, Santry

REFERENCES:
- [Result] Maheshwari AV, Blum YC, Shekhar L, Ranawat AS, Ranawat CS. Multimodal pain management after total hip and knee arthroplasty at the Ranawat Orthopaedic Center. Clin Orthop Relat Res. 2009 Jun;467(6):1418-23. doi: 10.1007/s11999-009-0728-7. Epub 2009 Feb 13. PMID 19214642
- [Result] Parvataneni HK, Shah VP, Howard H, Cole N, Ranawat AS, Ranawat CS. Controlling pain after total hip and knee arthroplasty using a multimodal protocol with local periarticular injections: a prospective randomized study. J Arthroplasty. 2007 Sep;22(6 Suppl 2):33-8. doi: 10.1016/j.arth.2007.03.034. Epub 2007 Jul 26. PMID 17823012
- [Result] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Result] Essving P, Axelsson K, Kjellberg J, Wallgren O, Gupta A, Lundin A. Reduced hospital stay, morphine consumption, and pain intensity with local infiltration analgesia after unicompartmental knee arthroplasty. Acta Orthop. 2009 Apr;80(2):213-9. doi: 10.3109/17453670902930008. PMID 19404806
- [Result] Fu P, Wu Y, Wu H, Li X, Qian Q, Zhu Y. Efficacy of intra-articular cocktail analgesic injection in total knee arthroplasty - a randomized controlled trial. Knee. 2009 Aug;16(4):280-4. doi: 10.1016/j.knee.2008.12.012. Epub 2009 Mar 18. PMID 19299145
- [Result] Lombardi AV Jr, Berend KR, Mallory TH, Dodds KL, Adams JB. Soft tissue and intra-articular injection of bupivacaine, epinephrine, and morphine has a beneficial effect after total knee arthroplasty. Clin Orthop Relat Res. 2004 Nov;(428):125-30. doi: 10.1097/01.blo.0000147701.24029.cc. PMID 15534532
- [Result] Nechleba J, Rogers V, Cortina G, Cooney T. Continuous intra-articular infusion of bupivacaine for postoperative pain following total knee arthroplasty. J Knee Surg. 2005 Jul;18(3):197-202. doi: 10.1055/s-0030-1248181. PMID 16152868
- [Result] Toftdahl K, Nikolajsen L, Haraldsted V, Madsen F, Tonnesen EK, Soballe K. Comparison of peri- and intraarticular analgesia with femoral nerve block after total knee arthroplasty: a randomized clinical trial. Acta Orthop. 2007 Apr;78(2):172-9. doi: 10.1080/17453670710013645. PMID 17464603
- [Result] Andersen KV, Pfeiffer-Jensen M, Haraldsted V, Soballe K. Reduced hospital stay and narcotic consumption, and improved mobilization with local and intraarticular infiltration after hip arthroplasty: a randomized clinical trial of an intraarticular technique versus epidural infusion in 80 patients. Acta Orthop. 2007 Apr;78(2):180-6. doi: 10.1080/17453670710013654. PMID 17464604
- [Result] Andersen LJ, Poulsen T, Krogh B, Nielsen T. Postoperative analgesia in total hip arthroplasty: a randomized double-blinded, placebo-controlled study on peroperative and postoperative ropivacaine, ketorolac, and adrenaline wound infiltration. Acta Orthop. 2007 Apr;78(2):187-92. doi: 10.1080/17453670710013663. PMID 17464605
- [Result] Chen DW, Hsieh PH, Huang KC, Hu CC, Chang YH, Lee MS. Continuous intra-articular infusion of bupivacaine for post-operative pain relief after total hip arthroplasty: a randomized, placebo-controlled, double-blind study. Eur J Pain. 2010 May;14(5):529-34. doi: 10.1016/j.ejpain.2009.08.008. Epub 2009 Sep 24. PMID 19781964
- [Result] Fischer HB, Simanski CJ. A procedure-specific systematic review and consensus recommendations for analgesia after total hip replacement. Anaesthesia. 2005 Dec;60(12):1189-202. doi: 10.1111/j.1365-2044.2005.04382.x. PMID 16288617
- [Result] Foster RH, Markham A. Levobupivacaine: a review of its pharmacology and use as a local anaesthetic. Drugs. 2000 Mar;59(3):551-79. doi: 10.2165/00003495-200059030-00013. PMID 10776835
- [Result] Gristwood RW, Greaves JL. Levobupivacaine: a new safer long acting local anaesthetic agent. Expert Opin Investig Drugs. 1999 Jun;8(6):861-76. doi: 10.1517/13543784.8.6.861. PMID 15992136
- [Result] Gwilym SE, Pollard TC, Carr AJ. Understanding pain in osteoarthritis. J Bone Joint Surg Br. 2008 Mar;90(3):280-7. doi: 10.1302/0301-620X.90B3.20167. PMID 18310746
- [Result] Gallagher EJ, Bijur PE, Latimer C, Silver W. Reliability and validity of a visual analog scale for acute abdominal pain in the ED. Am J Emerg Med. 2002 Jul;20(4):287-90. doi: 10.1053/ajem.2002.33778. PMID 12098173